CLINICAL TRIAL: NCT07239206
Title: Effectiveness of Serious Game on Facilitating Targeted Temperature Management Knowledge and Situational Awareness Among Critical Care Nurses
Brief Title: Serious Game for Improving Targeted Temperature Management Knowledge and Situational Awareness in Critical Care Nurses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Clinical Trial Center (Other)
Responsible Party: Sponsor-Investigator, National Taiwan University Clinical Trial Center, National Taiwan University Hospital, National Taiwan University Hospital
Organization: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202507084RINA
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Targeted Temperature Management; Nursing Education; Serious Game; Cardiac Arrest
Keywords: Targeted temperature management; Serious game
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into two parallel groups. The experimental group will receive lecture-based teaching combined with a digital serious game intervention, while the control group will receive lecture-based teaching with case discussion only. Randomization will be performed at the beginning of each class session to ensure balanced group allocation.
Who Masked: Participant
Masking Description: Participants are blinded to group assignment until the intervention begins. Investigators are aware of allocation to deliver the assigned teaching method.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Serious Game + Lecture (Experimental): Participants in this arm will receive lecture-based teaching combined with a digital serious game designed to enhance targeted temperature management (TTM) knowledge and situational awareness. The serious game includes interactive case scenarios, decision-making tasks, and real-time feedback to simulate ICU situations and reinforce learning.
  Interventions: Behavioral: Serious Game Intervention; Behavioral: Lecture-based Education
- Active Comparator: Lecture Only (Active Comparator): Participants in this arm will receive lecture-based teaching with case discussion only, covering the same targeted temperature management (TTM) content as the experimental group. No serious game intervention will be provided.
  Interventions: Behavioral: Lecture-based Education

INTERVENTIONS:
Behavioral: Serious Game Intervention — A digital serious game designed to train critical care nurses in targeted temperature management (TTM). The game features case-based simulations, interactive decision-making, and real-time feedback to improve clinical reasoning and situational awareness.
  Arms: Experimental: Serious Game + Lecture
Behavioral: Lecture-based Education — Standard lecture-based teaching covering the principles, procedures, and nursing care of targeted temperature management (TTM). Participants in this group do not receive the serious game component.

SUMMARY:
This randomized controlled trial aims to evaluate the effectiveness of a serious game in improving targeted temperature management (TTM) knowledge and situational awareness among critical care nurses. A total of 120 nurses from adult intensive care units will be randomly assigned to either a control group receiving traditional lecture-based teaching or an experimental group receiving lecture-based teaching combined with a digital serious game. Outcomes will be measured using a TTM knowledge test, a situational awareness scale, and a system usability scale. The findings will provide evidence for the use of serious games as an innovative educational strategy to enhance post-resuscitation care quality and patient safety.

DETAILED DESCRIPTION:
Targeted temperature management (TTM) is an evidence-based neuroprotective strategy recommended for patients resuscitated after cardiac arrest. Despite its clinical importance, critical care nurses often lack sufficient knowledge and situational awareness to effectively implement TTM, due to limited exposure to relevant cases and time constraints in training. Conventional teaching methods, while beneficial, face challenges such as limited resources, time, and opportunities for repeated practice.

Serious games, which integrate educational content with interactive digital game elements, offer a flexible and engaging learning tool that enables repeated practice in a safe, simulated environment. Previous studies have shown that serious games can enhance learners' motivation, knowledge retention, and decision-making skills.

This study will develop and implement a serious game specifically designed for TTM education. The randomized controlled trial will enroll 120 intensive care unit nurses, randomly allocated into two groups: the control group will receive lecture-based teaching with case discussion, while the experimental group will receive the same content supplemented with the serious game for additional practice. All participants will complete a pre-test, a post-test one week after the intervention, and a follow-up test at six weeks.

The primary outcome will be the improvement in TTM knowledge, and secondary outcomes will include situational awareness and system usability (experimental group only). The study is expected to provide evidence that serious games are an effective and scalable strategy for enhancing TTM-related knowledge and situational awareness, thereby supporting better quality of post-resuscitation care and patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Registered nurses currently working in adult intensive care units (medical, surgical, or mixed ICUs).
* Able to read and understand Chinese.
* Willing to participate and provide informed consent.
* Available to complete pre-test, post-test, and follow-up assessments.

Exclusion Criteria:

* Nurses working in pediatric or neonatal ICUs.
* Nurses holding administrative or supervisory positions (non-clinical).
* Nurses currently participating in other TTM-related educational or research programs.
* Individuals unable to complete the intervention or evaluation schedule.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Targeted Temperature Management (TTM) Knowledge Score | Baseline (pre-test), 1 week after intervention, and 6 weeks after intervention
  TTM knowledge will be assessed using a validated 16-item multiple-choice questionnaire developed based on current clinical guidelines. Scores range from 0 to 100, with higher scores indicating greater knowledge of targeted temperature management principles and nursing care.
Change in Situational Awareness (SA) Score | Baseline, 1 week after intervention, and 6 weeks after intervention
  Situational awareness will be measured using a 11-item Likert scale (1-5) questionnaire assessing perception, comprehension, and projection dimensions. Total scores range from 12 to 60, with higher scores indicating greater situational awareness in clinical TTM scenarios.
System Usability Scale (SUS) Score | 1 week after intervention (experimental group only)
  The usability of the serious game will be evaluated using the 10-item System Usability Scale (SUS). Scores range from 0 to 100, with higher scores indicating better system usability and learner satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nolan JP, Morley PT, Vanden Hoek TL, Hickey RW, Kloeck WG, Billi J, Bottiger BW, Morley PT, Nolan JP, Okada K, Reyes C, Shuster M, Steen PA, Weil MH, Wenzel V, Hickey RW, Carli P, Vanden Hoek TL, Atkins D; International Liaison Committee on Resuscitation. Therapeutic hypothermia after cardiac arrest: an advisory statement by the advanced life support task force of the International Liaison Committee on Resuscitation. Circulation. 2003 Jul 8;108(1):118-21. doi: 10.1161/01.CIR.0000079019.02601.90. No abstract available. PMID 12847056
- [Background] Gorbanev I, Agudelo-Londono S, Gonzalez RA, Cortes A, Pomares A, Delgadillo V, Yepes FJ, Munoz O. A systematic review of serious games in medical education: quality of evidence and pedagogical strategy. Med Educ Online. 2018 Dec;23(1):1438718. doi: 10.1080/10872981.2018.1438718. PMID 29457760
- [Background] Nolan JP, Sandroni C, Bottiger BW, Cariou A, Cronberg T, Friberg H, Genbrugge C, Haywood K, Lilja G, Moulaert VRM, Nikolaou N, Olasveengen TM, Skrifvars MB, Taccone F, Soar J. European Resuscitation Council and European Society of Intensive Care Medicine guidelines 2021: post-resuscitation care. Intensive Care Med. 2021 Apr;47(4):369-421. doi: 10.1007/s00134-021-06368-4. Epub 2021 Mar 25. PMID 33765189